CLINICAL TRIAL: NCT00753558
Title: A Randomized,Double-Blind,Placebo-Controled Trial of Selective Digestive Decontamination Using Oral Gentamicin and Oral Polymyxin E for Eradication of Carbapenem-Resistant Klebsiella Pneumoniae Carriage
Brief Title: Selective Digestive Decontamination in Carriers of Carbapenem-resistant Klebsiella Pneumoniae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Other Study IDs: sor475808CTIL
Record Dates: First submitted 2008-09-02; First posted 2008-09-16 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Carriage of Carbapemen-resistant Klebsialle Pneumoniae

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): Oral solution of 0.45% saline and oral solution of H2O & saccharine. Oral gel composed of mineral oil, gelatine powder, pectin, sodium carboxymethylcellulose, polyethylene
  Interventions: Drug: Arm #1 :Oral solution and buccal gel of gentamicin and polymyxin E. Arm #2: Placebo.
- 1 (Active Comparator): Oral solution and buccal gel of gentamicin and polymyxin E
  Interventions: Drug: Arm #1 :Oral solution and buccal gel of gentamicin and polymyxin E. Arm #2: Placebo.

INTERVENTIONS:
Drug: Arm #1 :Oral solution and buccal gel of gentamicin and polymyxin E. Arm #2: Placebo. — Arm #1: Oral gentamicin & polymyxin E, gentamicin & polymyxin E buccal gel.
  Arm #2: Oral placebo solutions, placebo buccal gel.

SUMMARY:
There is an urgent need to control our current national outbreak of carbapenem-resistant Klebsiella pneumoniae (CRKP). The purpose of this study is to eradicate CRKP gastrointestinal carriage using selective digestive decontamination (SDD); with buccal and oral gentamicin and polymyxin E administration. This will reduce infections and hopefully mortality caused by CRKP.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized men and women with a positive rectal swab for CRKP
* Age 18 years or older

Exclusion Criteria:

* Age less than 18 years
* Pregnant women, lactating women
* A known allergy to the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2008-11; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Eradication of CRKP carriage measured by negative rectal swabs | Two days after treatment ends

SECONDARY OUTCOMES:
No new in-hospital acquisition of CRKP | Six weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

REFERENCES:
- [Background] Silvestri L, van Saene HK, Milanese M, Gregori D, Gullo A. Selective decontamination of the digestive tract reduces bacterial bloodstream infection and mortality in critically ill patients. Systematic review of randomized, controlled trials. J Hosp Infect. 2007 Mar;65(3):187-203. doi: 10.1016/j.jhin.2006.10.014. Epub 2007 Jan 22. PMID 17244516
- [Background] van Saene HK, Petros AJ, Ramsay G, Baxby D. All great truths are iconoclastic: selective decontamination of the digestive tract moves from heresy to level 1 truth. Intensive Care Med. 2003 May;29(5):677-90. doi: 10.1007/s00134-003-1722-2. Epub 2003 Apr 10. PMID 12687326
- [Background] Agusti C, Pujol M, Argerich MJ, Ayats J, Badia M, Dominguez MA, Corbella X, Ariza J. Short-term effect of the application of selective decontamination of the digestive tract on different body site reservoir ICU patients colonized by multi-resistant Acinetobacter baumannii. J Antimicrob Chemother. 2002 Jan;49(1):205-8. doi: 10.1093/jac/49.1.205. PMID 11751791
- [Background] Silvestri L, Mannucci F, van Saene HK. Selective decontamination of the digestive tract: a life saver. J Hosp Infect. 2000 Jul;45(3):185-90. doi: 10.1053/jhin.2000.0737. PMID 10896796
- [Background] de Jonge E, Schultz MJ, Spanjaard L, Bossuyt PM, Vroom MB, Dankert J, Kesecioglu J. Effects of selective decontamination of digestive tract on mortality and acquisition of resistant bacteria in intensive care: a randomised controlled trial. Lancet. 2003 Sep 27;362(9389):1011-6. doi: 10.1016/S0140-6736(03)14409-1. PMID 14522530
- [Background] Leone M, Albanese J, Antonini F, Nguyen-Michel A, Martin C. Long-term (6-year) effect of selective digestive decontamination on antimicrobial resistance in intensive care, multiple-trauma patients. Crit Care Med. 2003 Aug;31(8):2090-5. doi: 10.1097/01.CCM.0000079606.16776.C5. PMID 12973164
- [Result] Brun-Buisson C, Legrand P, Rauss A, Richard C, Montravers F, Besbes M, Meakins JL, Soussy CJ, Lemaire F. Intestinal decontamination for control of nosocomial multiresistant gram-negative bacilli. Study of an outbreak in an intensive care unit. Ann Intern Med. 1989 Jun 1;110(11):873-81. doi: 10.7326/0003-4819-110-11-873. PMID 2655521